CLINICAL TRIAL: NCT04964193
Title: Bioequivalence Study of 2 mg Cyproterone Acetate and 0.035 mg Ethinyl Estradiol in Indonesian Healthy Females
Brief Title: Bioequivalence Study of Cyproterone Acetate and Ethinyl Estradiol in Healthy Female Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PT Sydna Farma (Industry)
Collaborators: PT Pharma Metric Labs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 440/STD/PML/2018
Record Dates: First submitted 2021-04-14; First posted 2021-07-16 (Actual); Results first posted 2022-01-31 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: Drug Use
Keywords: cyproterone acetate; ethinyl estradiol; bioequivalence; cross-over design study; pharmacokinetics; Indonesian healthy female
MeSH Terms: interventions — Cyproterone Acetate; Ethinyl Estradiol

STUDY DESIGN:
Intervention Model Description: Randomized, single blind, two-period, single dose, crossover study with three weeks washout period in 24 healthy female subjects under fasting condition.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elzsa film-coated tablet (Experimental): Participants received Elzsa film-coated tablet (2 mg cyproterone acetate + 0.035 mg ethinylestradiol) with 240 mL of water
  Interventions: Drug: Elzsa film-coated tablet
- Diane-35 Sugar-coated tablet (Active Comparator): Participants received Diane-35 Sugar-coated tablet ( 2 mg cyproterone acetate + 0.035 mg ethinylestradiol) with 240 mL of water
  Interventions: Drug: Diane-35 Sugar-coated tablet

INTERVENTIONS:
Drug: Elzsa film-coated tablet — Administered with 240 mL of water
  Other Names: 2 mg cyproterone acetate + 0.035 mg ethinylestradiol
  Arms: Elzsa film-coated tablet
Drug: Diane-35 Sugar-coated tablet — Administered with 240 mL of water
  Other Names: 2 mg cyproterone acetate + 0.035 mg ethinylestradiol
  Arms: Diane-35 Sugar-coated tablet

SUMMARY:
The study was conducted to investigate whether 2 mg cyproterone acetate (CPA) and 0.035 mg ethinyl estradiol (EE) film-coated tablet (Elzsa®) manufactured by PT. Sydna Farma was bioequivalent to its reference product, Diane®-35 sugar-coated tablet manufactured by Bayer Weimar GmbH, Germany, imported by PT. Bayer Indonesia, Depok, Indonesia.

DETAILED DESCRIPTION:
Twenty four healty female subjects were given a single dose of Elzsa® FCT or or Diane®-35 with 240 mL of water. Then the blood samples for CPA and EE were drawn and analyzed using LCMS/MS. All subjects sample plasma were analyzed for pharmacokinetic evaluation

ELIGIBILITY:
Inclusion criteria

The inclusion criteria are healthy female subjects who/with:

* have read the subject information and signed informed consent documents
* age 18 - 55 years
* body mass index between 18-25 kg/m2
* have a normal electrocardiogram
* blood pressure within normal range (90-120 mmHg for systolic blood pressure and 60-80 mmHg for diastolic blood pressure)
* heart rate within normal range (60-100 bpm)
* with absence of significant disease or clinically significant abnormal laboratory values on laboratory evaluation, medical history or physical examination during screening
* pass hormone screening related to cyproterone acetate and ethinyl estradiol

Exclusion criteria

Any of the following criteria will exclude the subject from the study:

* those who are pregnant and/or nursing woman.
* those with history of hypersensitivity to cyproterone acetate and ethinyl estradiol or other oral contraception or other ingredients in the drugs or a history of serious allergic reaction to any drug, significant allergic disease, allergic reaction, or active allergic.
* those with a history or presence medical condition which might significantly influence the pharmacokinetic of the study drug, e.g. chronic gastrointestinal disease, diarrhea, gastric surgery, renal insufficiency, hepatic dysfunction or cardiovascular disease.
* those with a history or presence of any coagulation disorder or clinically significant hematology abnormalities, thrombophlebitis, and thromboembolic disorder.
* those who are using any medication (prescription or non-prescription drug, food supplement, herbal medicine, oral contraception, anti-platelet drug), particularly the medication known to affect the pharmacokinetic of the study drug, within one week prior to the drug administration day.
* those who have participated in any clinical study within 3 months prior to the study (< 90 days).
* those who have donated or lost 300 ml (or more) of blood within 3 months prior to the study.
* those who smoke.
* those who are positive to HIV, HBsAg, and HCV tests (to be kept confidential).
* those with a history of drug or alcohol abuse within 12 months prior to screening for this study.
* those who are unlikely to comply with the protocol, e.g uncooperative attitude, inability to return for follow up visits, poor venous access.

Ages: 19 Years to 54 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2019-03-12 (Actual); Primary Completion 2019-07-04 (Actual); Study Completion 2019-09-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- PT Pharma Metric Labs, Multiple Locations, Jakarta Special Capital Region, Indonesia

REFERENCES:
- [Result] Luque-Ramirez M, Alvarez-Blasco F, Botella-Carretero JI, Martinez-Bermejo E, Lasuncion MA, Escobar-Morreale HF. Comparison of ethinyl-estradiol plus cyproterone acetate versus metformin effects on classic metabolic cardiovascular risk factors in women with the polycystic ovary syndrome. J Clin Endocrinol Metab. 2007 Jul;92(7):2453-61. doi: 10.1210/jc.2007-0282. Epub 2007 Apr 10. PMID 17426085
- [Result] Bhattacharya SM, Jha A. Comparative study of the therapeutic effects of oral contraceptive pills containing desogestrel, cyproterone acetate, and drospirenone in patients with polycystic ovary syndrome. Fertil Steril. 2012 Oct;98(4):1053-9. doi: 10.1016/j.fertnstert.2012.06.035. Epub 2012 Jul 13. PMID 22795636
- [Result] Elger W, Beier S, Pollow K, Garfield R, Shi SQ, Hillisch A. Conception and pharmacodynamic profile of drospirenone. Steroids. 2003 Nov;68(10-13):891-905. doi: 10.1016/j.steroids.2003.08.008. PMID 14667981
- [Result] Bitzer J, Romer T, Lopes da Silva Filho A. The use of cyproterone acetate/ethinyl estradiol in hyperandrogenic skin symptoms - a review. Eur J Contracept Reprod Health Care. 2017 Jun;22(3):172-182. doi: 10.1080/13625187.2017.1317339. Epub 2017 Apr 27. PMID 28447864
- [Result] Speck U, Wendt H, Schulze PE, Jentsch D. Bio-availability and pharmacokinetics of cyproterone acetate-14C and ethinyloestradiol-3H after oral administration as a coated tablet (SH B 209 AB). Contraception. 1976 Aug;14(2):151-63. doi: 10.1016/0010-7824(76)90083-4. PMID 949892
- [Result] Kuhnz W, Staks T, Jutting G. Pharmacokinetics of cyproterone acetate and ethinylestradiol in 15 women who received a combination oral contraceptive during three treatment cycles. Contraception. 1993 Dec;48(6):557-75. doi: 10.1016/0010-7824(93)90118-q. PMID 8131397
- [Result] Sedgwick P. Bias in randomised controlled trials: comparison of crossover group and parallel group designs. BMJ. 2015 Aug 7;351:h4283. doi: 10.1136/bmj.h4283. No abstract available. PMID 26253465
- [Result] Garcia R, Benet M, Arnau C, Cobo E. Efficiency of the cross-over design: an empirical estimation. Stat Med. 2004 Dec 30;23(24):3773-80. doi: 10.1002/sim.2072. PMID 15580599
- [Result] Sedgwick P. What is a crossover trial? BMJ. 2014 May 9;348:g3191. doi: 10.1136/bmj.g3191. No abstract available. PMID 25134118
- [Result] Sedgwick P. Randomised controlled trials: "within subject" versus "between subject" designs. BMJ. 2014 Oct 24;349:g6435. doi: 10.1136/bmj.g6435. No abstract available. PMID 25954990
- See also: (accessed on Sep 18, 2020) — http://www.ema.europa.eu/en/documents/referral/cyproterone/ethinylestradiol-containing-medicines-article-107i-procedure-prac-assessment-report_en.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Test Drug First, Then Reference Drug: New (test) Elzsa film-coated tablet (2 mg cyproterone acetate + 0.035 mg ethinylestradiol) as a single oral dose in the first intervention period, and marketed (reference) Diane®-35 sugar-coated tablet (2 mg cyproterone acetate + 0.035 mg ethinylestradiol) as a single oral dose in the second intervention period (after washout period).
- Diane-35 Sugar-coated Tablet: Marketed (reference) Diane-35 Sugar-coated tablet (2 mg cyproterone acetate + 0.035 mg ethinylestradiol) as a single oral dose in the first intervention period, and new (test) Elzsa film-coated tablet (2 mg cyproterone acetate + 0.035 mg ethinylestradiol) as a single oral dose in the second intervention period (after washout period).
Period: 1st Intervention
Arm/Group | Test Drug First, Then Reference Drug | Diane-35 Sugar-coated Tablet
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Washout = Three Weeks
Arm/Group | Test Drug First, Then Reference Drug | Diane-35 Sugar-coated Tablet
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: 2nd Intervention
Arm/Group | Test Drug First, Then Reference Drug | Diane-35 Sugar-coated Tablet
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Number of Participants: All participants received 2 mg cyproterone acetate + 0.035 mg ethinylestradiol tablet (new and marketed)
Arm/Group | Total Number of Participants
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics Parameter
Description: Maximum plasma concentration (Cmax)
Time Frame: before dosing (0 h) and at 15, 30, 45 min, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 15, 24, 36, 48 and 72 hours after dosing
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Elzsa Film-coated Tablet | Diane-35 Sugar-coated Tablet
Number analyzed (Participants) | 24 | 24
pg/mL
  Cmax of Cyproterone Acetate | 17.39 (13.77) | 16.20 (13.81)
  Cmax of Ethinyl Estradiol | 103.69 (47.42) | 93.61 (47.16)

2. Primary Outcome: Pharmacokinetics Parameter
Description: Area Under Curve from 0 to 72 hours (AUCt)
Time Frame: before dosing (0 h) and at 15, 30, 45 min, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 15, 24, 36, 48 and 72 hours after dosing
Measure: Mean (Standard Deviation); unit: pg*hr/mL
Arm/Group | Elzsa Film-coated Tablet | Diane-35 Sugar-coated Tablet
Number analyzed (Participants) | 24 | 24
pg*hr/mL
  AUC0-t of Cyproterone Acetate | 132.56 (73.19) | 127.54 (89.41)
  AUC0-t of Ethinyl Estradiol | 870.45 (383.56) | 842.56 (398.66)

ADVERSE EVENTS:
Time Frame: at 15, 30, 45 min, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 9, 15, 24, 36, 48 and 72 hours after dosing
Description: [Not Specified]
Groups:
- Elzsa Film-coated Tablet: New (test) Elzsa film-coated tablet (2 mg cyproterone acetate + 0.035 mg ethinylestradiol) as a single oral dose.
- Diane-35 Sugar-coated Tablet: Marketed (reference) Diane-35 Sugar-coated tablet ( 2 mg cyproterone acetate + 0.035 mg ethinylestradiol) as a single oral dose.
Arm/Group | Elzsa Film-coated Tablet | Diane-35 Sugar-coated Tablet
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 6/24 | 9/24
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Elzsa Film-coated Tablet (N=24) | Diane-35 Sugar-coated Tablet (N=24)
Dizziness (General disorders) | 1 (1) | 2 (2)
Drowsiness (General disorders) | 1 (1) | 1 (1)
Headache (General disorders) | 1 (1) | 2 (2)
Breast tenderness or Breast discomfort (Reproductive system and breast disorders) | 1 (1) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Toothache (General disorders) | 1 (1) | 0 (0)
Pharyngitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Frequently Urination (Renal and urinary disorders) | 0 (0) | 1 (1)
Syncope (General disorders) | 1 (1) | 0 (0)
Flu like symptoms (Runny rose nose, headache) (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-12): https://cdn.clinicaltrials.gov/large-docs/93/NCT04964193/Prot_SAP_001.pdf